CLINICAL TRIAL: NCT05861258
Title: Pharmacokinetic Study of Minocycline in Patients With Pulmonary Nontuberculous Mycobacterial Disease
Acronym: Mino-PK
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial was terminated prematurely after the enrollment of 12 out of 15 planned subjects, due to a lack of personnel and no option to continue study measurements.
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL69313.091.19
Record Dates: First submitted 2023-05-04; First posted 2023-05-16 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2024-11

CONDITIONS: Mycobacterium Avium Complex Pulmonary Disease
Keywords: Pharmacokinetics; Minocycline; Rifampicin
MeSH Terms: conditions — cyclopia sequence | interventions — Minocycline

STUDY DESIGN:
Intervention Model Description: A single group, two-period, fixed-order pharmacokinetic study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Minocycline — Patients with M. avium complex pulmonary disease will receive 200 mg of minocycline for 5 days before starting rifampicin and after 1 month (±1 week) of receiving rifampicin. Antimycobacterial drugs other than rifampicin can be started prior to or simultaneous with the first minocycline dosing period as part of standard care. At day 5 of both minocycline dosing periods, blood will be sampled for minocycline plasma concentration measurements at T = 0, 1, 2, 3, 4, 6, 8 and 24 hours.

SUMMARY:
Antimycobacterial treatment of M. avium complex pulmonary disease (MAC-PD) has suboptimal cure rates and is challenging due to frequent adverse drug reactions and drug-drug interactions. Hence, there is an urgent need for improved treatment regimens with effective and tolerable antibiotics.

Minocycline is a well-tolerated, orally administered tetracycline-type antibiotic with in vitro activity against MAC, but pharmacokinetic data in the target population is lacking. Moreover, rifampicin, a strong inducer of cytochrome P450 enzymes involved in drug metabolism and of various drug transporters, is part of the current first-line MAC-PD treatment regimen and has a substantial interaction with doxycycline, a related tetracycline.

Pharmacokinetic data in the target population will allow us to propose an appropriate dose of minocycline when co-administered with or without rifampicin

Mino-PK is an open label, one-arm, two-period, fixed-order pharmacokinetic study that will assess exposure to minocycline in MAC-PD patients with and without concurrent use of rifampicin. Subjects will receive two 5-day dosing periods of minocycline; the first without and second with concurrent use of rifampicin. Minocycline plasma concentrations will be determined after both dosing periods.

ELIGIBILITY:
Inclusion Criteria:

* 2020 guideline (ATS/ERS/ESCMID/IDSA) diagnostic criteria for nontuberculous mycobacterial pulmonary disease are met, i.e. the patient is symptomatic, has nodules, bronchiectasis or fibro-cavitary lesions seen on (HR)CT scan of the lungs and ≥2 positive sputum cultures or one positive bronchoalveolar lavage culture of the same M. avium complex species.
* At least one of the positive cultures must be done in the last 4 months before inclusion.
* The subject is eligible to start the guideline-recommended rifampicin-based regimen according to the treating physician.
* Age ≥ 18 years.
* Signed and dated patient informed consent.

Exclusion Criteria:

* A relevant medical history or current condition that might interfere with drug absorption, distribution, metabolism or excretion (i.e. chronic gastro-intestinal disease, renal or hepatic disease).
* Diagnosed with cystic fibrosis (as this may affect the pharmacokinetics of drugs).
* Pregnant or breastfeeding (contra-indications for minocycline) or inadequate contraceptive measures (in view of the administration of rifampicin which interacts with oral contraceptive drugs, adequate contraceptive measures are abstinence from sexual activities and barrier methods).
* Use of drugs that cause a relevant drug interaction with minocycline, i.e. oral magnesium, , bismuth, aluminium, calcium, zinc or iron containing formulations, antacid drugs and drugs besides rifampicin that are strong inducers of metabolic enzymes, including barbiturates, carbamazepin and phenytoin (as judged by the investigators).
* ALAT > 3 times the upper limit of normal (normal <45 U/l).
* ASAT > 3 times the upper limit of normal (normal <35 U/l).
* An abnormal serum creatinine level (defined as a level that is higher than the upper limit of normal, i.e. >110 umol/l).
* Active alcohol abuse.
* Hypersensitivity to minocycline or to other tetracycline antibiotics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-05-08 (Actual); Primary Completion 2025-05-14 (Actual); Study Completion 2025-06-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters of minocycline in MAC-PD patients without concurrent use of rifampicin. | Day 5 of the first minocycline dosing period
  The area under the curve (AUC0-24h)
Pharmacokinetic parameters of minocycline in MAC-PD patients without concurrent use of rifampicin. | Day 5 of the first minocycline dosing period
  The peak plasma concentration (Cmax)
Pharmacokinetic parameters of minocycline in MAC-PD patients without concurrent use of rifampicin. | Day 5 of the first minocycline dosing period
  The plasma trough concentration (Cmin)

SECONDARY OUTCOMES:
Pharmacokinetic parameters of minocycline in MAC-PD patients with concurrent use of rifampicin. | Day 5 of the second minocycline dosing period
  The area under the curve (AUC0-24h)
Pharmacokinetic parameters of minocycline in MAC-PD patients with concurrent use of rifampicin. | Day 5 of the second minocycline dosing period
  The peak plasma concentration (Cmax)
Pharmacokinetic parameters of minocycline in MAC-PD patients with concurrent use of rifampicin. | Day 5 of the second minocycline dosing period
  The plasma trough concentration (Cmin)
Pharmacokinetic parameters of rifampicin in MAC-PD patients | Day 5 of the second minocycline dosing period
  The peak plasma concentration (Cmax)
Adverse Events | Through study completion, an average of 6 weeks
  The number of (participants with) adverse events will be measured. Adverse events will be graded according to the 'Common Terminology Criteria for Adverse Events' (CTCAE)

CONTACTS AND LOCATIONS:
Overall Officials: Wouter Hoefsloot, MSc, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Medical Center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The pseudonymized participant data will be accessible in the Radboud Data Repository under restricted access, only if the participant has provided consent. Requests for access will be checked, by a data access committee (DAC) formed by the sponsor (i.e. PI and other research members / coordinators)
  The following data will be shared:
  * Final versions of data used for analysis
  * Documentation/codebooks necessary for understanding the data
  * The .xml file that contains the full structure of the eCRF build in Castor EDC
  * Read me.txt for understanding the structure and content of the documents
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will become available for 15 years after the first study report has been published.
Access Criteria: To be determined
URL: https://data.ru.nl/?0

REFERENCES:
- [Background] Daley CL, Iaccarino JM, Lange C, Cambau E, Wallace RJ Jr, Andrejak C, Bottger EC, Brozek J, Griffith DE, Guglielmetti L, Huitt GA, Knight SL, Leitman P, Marras TK, Olivier KN, Santin M, Stout JE, Tortoli E, van Ingen J, Wagner D, Winthrop KL. Treatment of nontuberculous mycobacterial pulmonary disease: an official ATS/ERS/ESCMID/IDSA clinical practice guideline. Eur Respir J. 2020 Jul 7;56(1):2000535. doi: 10.1183/13993003.00535-2020. Print 2020 Jul. PMID 32636299